CLINICAL TRIAL: NCT00198978
Title: Multicenter Study To Optimize Treatment in Elderly Patients (> 55 Years, No Upper Age Limit) With Acute Lymphoblastic Leukemia (GMALL Elderly 1/2003)(Amend 2)
Brief Title: German Multicenter Trial for Treatment of Elderly Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Head of GMALL, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL02
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Adult Acute Lymphocytic Leukemia
Keywords: ALL; Treatment; Elderly; De novo
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Dexamethasone; Prednisolone; Cytarabine; Idarubicin; Granulocyte Colony-Stimulating Factor; Mercaptopurine; Methotrexate; Rituximab; Vincristine; Asparaginase

ARMS (1):
- Interventional arm (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Dexamethasone / Prednisolone; Drug: Cytarabine; Drug: Idarubicin; Drug: Granulocyte-Colony-Stimulating Factor; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Rituximab; Drug: HDARAC; Drug: Vincristine; Drug: Depocyte; Drug: Asparaginase

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Dexamethasone / Prednisolone
Drug: Cytarabine
Drug: Idarubicin
Drug: Granulocyte-Colony-Stimulating Factor
Drug: Mercaptopurine
Drug: Methotrexate
Drug: Rituximab
Drug: HDARAC
Drug: Vincristine
Drug: Depocyte
Drug: Asparaginase

SUMMARY:
The study evaluates the efficacy and tolerability of a dose-reduced chemotherapy for the treatment of elderly patients with acute lymphoblastic leukemia. In patients with expression of CD20 on leukemic cells the efficacy and tolerability of additional application of Rituximab together with chemotherapy is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia (pro B, pre B, c-ALL or T-ALL), proved by morphology and immunophenotyping
* Age > 55 yrs (no upper age limit)
* Written informed consent

Exclusion Criteria:

* Severe leukemia associated complications, not controllable before therapy onset e.g.
* life threatening infections as sepsis, pneumonia, hypoxia, shock, life threatening bleeding)
* Severe comorbidity e.g.
* decompensated renal failure if not caused by leukemia with Creatinine > 2x ULN
* heart failure (NYHA II/IV), instable Angina, significant coronary stenosis
* hepatic insufficiency e.g. liver cirrhosis or chronic active hepatitis with bilirubin > 1,5 x ULN and/or ASA, ALA, AP > 2,5 ULN
* decompensated metabolic disturbances (e.g. not controllable diabetes)
* severe obstructive or restrictive pulmonary disease with hypoxaemia
* Severe psychiatric illness or other circumstances which may compromise cooperation of the patient
* Active second neoplasia
* HIV infection
* Severely reduced general condition
* Cytostatic pre-treatment of ALL
* Chemotherapy treatment of any other malignancy during the last 5 years
* Participation in other clinical trials interfering with the study therapy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Remission rate (cytologic, molecular) | After induction; approximately 6 wks (exact time frame not specified)
Toxicity (CTC) | After each cycle; time-frame not specified
Survival time, Duration of Remission | at 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD,PhD, Study Chair — University of Frankfurt, Medical Dept. II
Locations (1):
- University of Frankfurt, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- [Derived] Topp MS, Gokbuget N, Zugmaier G, Degenhard E, Goebeler ME, Klinger M, Neumann SA, Horst HA, Raff T, Viardot A, Stelljes M, Schaich M, Kohne-Volland R, Bruggemann M, Ottmann OG, Burmeister T, Baeuerle PA, Nagorsen D, Schmidt M, Einsele H, Riethmuller G, Kneba M, Hoelzer D, Kufer P, Bargou RC. Long-term follow-up of hematologic relapse-free survival in a phase 2 study of blinatumomab in patients with MRD in B-lineage ALL. Blood. 2012 Dec 20;120(26):5185-7. doi: 10.1182/blood-2012-07-441030. Epub 2012 Sep 28. PMID 23024237